CLINICAL TRIAL: NCT00861965
Title: A Phase I/II Study of Polyclonally Activated, Intentionally Mis-Matched, Allogeneic Th1 Memory Cells (AlloStimTM) in Patients With Relapsed or Refractory Hematological Malignancy Without Prior Conditioning
Brief Title: Bioengineered Allogeneic Immune Cells (AlloStim) Not Requiring HLA Donor Match for Blood Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: withdrawn due to poor recruitment
Sponsor: Mirror Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITL-001-HM
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2015-04

CONDITIONS: Advanced or Refractory Leukemia, Lymphoma, Multiple Myeloma
Keywords: Leukemia; Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): AlloStim-8
  Interventions: Biological: AlloStim-8

INTERVENTIONS:
Biological: AlloStim-8 — intravenous infusion of mis-matched AlloStim-8
Biological: AlloStim-8 — intravenous infusion of AlloStim-8 on day 7
Biological: AlloStim-8 — intravenous infusion of AlloStim-8 on day 14
Biological: AlloStim-8 — intravenous infusion of AlloStim-8 on day 21

SUMMARY:
This phase I/II clinical investigation is designed to determine the safety and anti-tumor effects of intravenous administration of the experimental immunotherapy drug, called AlloStim. The active ingredient of AlloStim is living, human immune cells that have been differentiated and expanded outside the body. Because AlloStim does not require HLA match, it is being evaluated as an alternative to allogeneic bone marrow/stem cell transplantation.

DETAILED DESCRIPTION:
AlloStim is being tested to determine if it might elicit the same anti-tumor mechanism that occurs in allogeneic bone marrow/stem cell transplant (BMT) procedures, without the toxicity associated with graft vs. host disease (GVHD). In allogeneic BMT settings, patients are first conditioned to weaken the immune system in order to enable the engraftment of allogeneic donor cells. Patients require a matched-tissue donor in this setting in order to enable engraftment and also to minimize GVHD toxicity. While allogeneic BMT is a potentially curatve therapy, the treatment-related mortality, mostly related to GVHD toxicity, is high. This toxicity limits the clinical utility of this procedure. AlloStim is being tested to determine if it might be a less toxic alternative to allogeneic BMT.

In this protocol, patients are not conditioned with chemotherapy prior to treatment. Therefore, the allogeneic cells in AlloStim are expected to be rejected by the patient's immune system within 24-48 hours of infusion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed hematological malignancy of 1 of the following types:

  * Acute Myeloid Leukemia (AML) meeting the following criteria:

    * Relapsed or primary refractory disease with ≤ 10% blasts in the peripheral blood and ≤ 20% blasts in the bone marrow.
  * Acute Lymphoblastic Leukemia (ALL) meeting the following criteria:

    * Relapsed or primarily refractory disease with ≤ 10% blasts in the peripheral blood and ≤ 20% blasts in the bone marrow
  * Chronic Myeloid Leukemia (CML)* with an inadequate response to imatinib meeting 1 of the following criteria:

    * Second or subsequent chronic phase
    * Accelerated phase [*Patients with CML in blast crisis (> 30% promyelocytes and myeloblasts in the bone marrow) are not eligible]
  * Non-Hodgkin's Lymphoma (NHL) including Mantle Cell Lymphoma (MCL) meeting 1 of the following criteria:

    * Primary refractory disease or in refractory relapse
    * Relapsed disease after autologous stem cell transplantation
    * Chemosensitive relapsed disease without CR to standard salvage therapy AND no option for autologous stem cell transplantation due to blood or marrow involvement or failure to harvest sufficient autologous stem cells.
  * Chronic Lymphocytic Leukemia (CLL) meeting both of the following criteria:

    * Stage III or IV disease
    * Refractory to fludarabine, Rituxan® and Campath® or refuses
  * Multiple Myeloma (MM) meeting 1 of the following criteria:

    * Primary refractory disease or in refractory relapse
    * Relapsed disease after autologous stem cell transplantation
  * Hodgkin's Disease

    * Relapsed after prior autologous transplant or after 2 or more combination chemotherapy regimens and ineligible for autologous stem cell transplant.
  * EBV driven lymphoproliferative disorders in immunocompetent patients progressing despite standard therapies, including:

    * T-cell Non-Hodgkin's Lymphoma
    * Burkitt's Lymphoma
    * EBV+ Hodgkin's Disease

      * Ability to comprehend the investigational nature of the study and provide informed consent.
      * Measurable or evaluable disease
      * Eastern Cooperative Oncology Group (ECOG) performance status of <2.
      * Age 18 years or older
      * Expected survival 6 months or longer
      * No radiation or chemotherapy in previous 2 weeks
      * No immunotherapy in the previous 4 weeks
      * Absence of active infection within 2 weeks
      * Adequate hepatic function, with total bilirubin level less than 1.2 times the upper limit of normal (ULN) and aspartate and alanine aminotransferase levels less than 2.5 times the ULN prior to infusion
      * Adequate bone marrow function defined as a white blood cell count of at least 2 x 109/L (2000/µL), absolute neutrophil count of at least 1 x 109/L (1000/µL), hemoglobin level of at least 80 g/L (8.0 g/dL), and a platelet count of at least 50 x 109/L (50,000/µL) priot to infusion. Patients who are transfusion- or growth factor-dependent are allowed, provided these values could be achieved with transfusion.
      * Adequate cardiovascular function defined as no ischemia, no new conduction system abnormalities, no class 3 or 4 New York Heart Association congestive heart failure, and no myocardial infarction in the previous 6 months. A ≥45% left ventricular ejection fraction (LVEF) required in the previous 6 months.
      * Adequate kidney function defined as serum creatinine level 1.5 mg/dL or less, or an estimated creatinine clearance level of at least 60 mL/min prior to infusion.
      * Adequate lung function defined as pulse oxymetry greater than or equal to 92% on room air prior to infusion, DLco≥50%, FEV1 and FVC ≥50% within 2 weeks
      * No known allergy to murine products or HAMA testing results within normal limits
      * No known allergy to bovine products

Exclusion Criteria:

* No pregnancy or breast feeding
* No known human immunodeficiency virus (HIV+)
* No seropositivity or active viral hepatitis (HBV+, HCV+)
* No prior allogeneic transplant (cell or organ)
* No serious concomitant medical or psychiatric conditions that could interfere with treatment.
* No EBV-induced lymphomas associated with immunosuppression, including patients with iatrogenic immunodeficiencies (such as organ transplant) or HIV-related immunodefiency.
* No chronic myelogenous leukemia in blast crisis.
* No myelodysplastic syndromes with refractory anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of administration of an intravenous AlloStim-9 infusion and to define any drug-related toxicity and reversibility of such toxicity | 7 days
evaluate the safety of administration of up to three consecutive daily intravenous AlloStim-8 booster infusions in patients that previously received a infusion of AlloStim-9 and to define any drug-related toxicity and reversibility of such toxicity | 90 days

SECONDARY OUTCOMES:
evaluate the anti-tumor effect of AlloStim infusions by evaluating the objective response rates | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michael Har-Noy, Study Director — Mirror Biologics, Inc.; Michael Berger, MD, Principal Investigator — Immunotherapy Clinical Associates, PC
Locations (1):
- Immunovative Clinical Research, Inc, Carlsbad, California, United States

REFERENCES:
- [Background] Har-Noy M, Zeira M, Weiss L, Fingerut E, Or R, Slavin S. Allogeneic CD3/CD28 cross-linked Th1 memory cells provide potent adjuvant effects for active immunotherapy of leukemia/lymphoma. Leuk Res. 2009 Apr;33(4):525-38. doi: 10.1016/j.leukres.2008.08.017. Epub 2008 Oct 1. PMID 18834631
- [Background] Har-Noy M, Zeira M, Weiss L, Slavin S. Completely mismatched allogeneic CD3/CD28 cross-linked Th1 memory cells elicit anti-leukemia effects in unconditioned hosts without GVHD toxicity. Leuk Res. 2008 Dec;32(12):1903-13. doi: 10.1016/j.leukres.2008.05.007. Epub 2008 Jun 18. PMID 18565579
- [Background] Har-Noy M, Slavin S. The anti-tumor effect of allogeneic bone marrow/stem cell transplant without graft vs. host disease toxicity and without a matched donor requirement? Med Hypotheses. 2008;70(6):1186-92. doi: 10.1016/j.mehy.2007.10.008. Epub 2007 Dec 3. PMID 18054441